CLINICAL TRIAL: NCT02805959
Title: Colonic Motility in Constipation and Aging: A Pilot Study With a New 3D Transit System
Brief Title: Colonic Motility in Constipation and Aging: A Study With a New 3D Transit System
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Fynne
Record Dates: First submitted 2016-05-04; First posted 2016-06-20 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-04

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Constipated, Elderly: Investigation with MTS for motility
  Interventions: Device: MTS2
- Constipation, Young: Investigation with MTS for motility
  Interventions: Device: MTS2
- Normal Bowel, Elderly: Investigation with MTS for motility
  Interventions: Device: MTS2
- Normal Bowel, Young: Investigation with MTS for motility
  Interventions: Device: MTS2

INTERVENTIONS:
Device: MTS2

SUMMARY:
To study the motility of the bowel in constipated patients. Looking at the difference between young and elderly patients with constipation.

ELIGIBILITY:
Inclusion Criteria:

* Constipation

Exclusion Criteria:

* Constipation caused by other disease

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with constipation
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Transit time through the small intestine and the colon. Both the total transit time, the regional transit times and the antegrade and retrograde movements are measured by the MTS system | The total transit time will differ between healthy and constipated but probably between 3-5 days.
  The measurements will all be at least three days long, but can be up to 5 days depending on the rate of bowel movements.

IPD SHARING:
Plan to Share IPD: No